CLINICAL TRIAL: NCT05453838
Title: Bioequivalence of a Diabetes Specific Tube Feed
Acronym: EQUIDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SBB22R&40700
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Postprandial Glucose Response

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New product - Original product (Other): All subjects will receive first product A and then product B. In addition, the reference product will also be received (three times a glucose solution during the trial).
  Interventions: Dietary Supplement: oral intake of one serving of the original and new product
- Original product - New product (Other): All subjects will receive first product B and then product A. In addition, the reference product will also be received (three times a glucose solution during the trial).
  Interventions: Dietary Supplement: oral intake of one serving of the original and new product

INTERVENTIONS:
Dietary Supplement: oral intake of one serving of the original and new product — 1) Intervention type: Dietary Supplement Intervention name: (visits 1, 3 and 5) Reference product Intervention description: Glucose solution 2) Intervention type: Dietary Supplement Intervention name: (visit 2 or 4) Diabetes specific tube feed Intervention description: : One serving new product 3) Intervention type: : Dietary Supplement Intervention name: (visit 2 or 4) Diabetes specific tube feed Intervention description: One serving original product

SUMMARY:
Nutricia has a range of nutritionally complete tube feeds on the market including some specific for diabetes patients. A new product is currently under development. The aim of the present study is to assess whether the postprandial glucose response of the new product is equivalent to the postprandial glucose response of an original product. In addition, the Glycaemic Index (GI) and Glycaemic Load (GL) of the adapted product will be determined. The study will have a crossover design with healthy volunteers taking one serving of both products in a randomized order. To determine GI and GL of the adapted product subjects will also receive a reference product. Subjects will visit the study site six times: one screening visit, three study visits to measure the glucose response to the reference product and two study visits to measure the glucose response to the test and control product.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 65 years
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 27.0 kg/m2
3. Written informed consent
4. Willingness and ability to comply with the protocol
5. Judged by the Investigator to be in good health

Exclusion Criteria:

1. Known Diabetes Mellitus type I or type II, rebound hypoglycaemia and/or any other medical condition that interferes with glucose metabolism
2. Any use of anticoagulants, systemic steroids, protease inhibitors or antipsychotics and/or any medication known to affect glucose tolerance and/or to influence digestion and absorption of nutrients within 1 week of screening, in opinion of the Investigator
3. Any known disease which influences digestion and absorption of nutrients within 1 week of screening (in the opinion of the Investigator)
4. Allergy to soy and/or any other known relevant food allergy or intolerance in opinion of the Investigator
5. Adherence to a strict vegan diet
6. Adherence to a weight loss program
7. Picky/fussy eater (being very selective about what to eat) or eating disorder
8. Known pregnancy and/or lactation
9. Current smoking or stopped smoking for < 1 month prior to screening (except for incidental smoking of ≤ 3 cigarettes/cigars/pipes per week on average in the last month)
10. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women (on average during the last 6 months)
11. Drug or medicine abuse in opinion of the Investigator
12. Any known bleeding disorder
13. Active participation in any other clinical study with investigational or marketed products concomitantly or within 4 weeks before study visit 1, in the opinion of the Investigator
14. Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the Investigator
15. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
16. Employees of Nutricia Research and/or family members or relatives of employees

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Blood glucose - Product A versus Product B | 120 minutes
  Blood glucose iAUC0-120 [mmol/L*min] [mmol/L]
Blood glucose - Product A versus Product B | 120 minutes
  Blood glucose iCmax [mmol/L] [mmol/L]

SECONDARY OUTCOMES:
GI new product | 120 minutes
  GI = blood glucose iAUC0-120 [mmol/L] of new product / mean blood glucose iAUC0-120 [mmol/L] of reference product
GL new product | 120 minutes
  GL = GI * available carbohydrate/given amount of carbohydrate

CONTACTS AND LOCATIONS:
Overall Officials: Monique Visser, PhD, Principal Investigator — Nutricia Research
Locations (1):
- NCRU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No